CLINICAL TRIAL: NCT06027034
Title: Effectiveness of a Digital Health Application for Psoriasis: Randomized Controlled Trial
Brief Title: Effectiveness of a Digital Health Application for Psoriasis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University of Giessen (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Psoriasis RCT 2023
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online program for psoriasis (GAIA-PSO-01) + TAU (Experimental): Participants allocated to the intervention group will receive access to an online program for psoriasis (GAIA-PSO-01) in addition to treatment as usual (TAU).
  Interventions: Behavioral: Online program for psoriasis (GAIA-PSO-01)
- TAU (No Intervention): Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: Online program for psoriasis (GAIA-PSO-01) — The program to-be-tested (GAIA-PSO-01) is an interactive online program for independent use by users with psoriasis. It focuses on recognized treatment elements of cognitive behavioral therapy (CBT) and behavior change techniques.
  Arms: Online program for psoriasis (GAIA-PSO-01) + TAU

SUMMARY:
This clinical trial with 348 patients with psoriasis aims to investigate the effectiveness of a self-guided online program for patients with psoriasis.

Patients will be randomized and allocated in a 1:1 ratio to either an intervention group, in which they will receive 12-month-access to an online program for psoriasis in addition to treatment as usual (TAU, n = 174), or to a control group, in which they will receive only TAU (n = 174). TAU is defined as any therapy prescribed or recommended by the GP or specialists (e.g. dermatologist, psychiatrist), which may include topical therapy, phototherapy, pharmacotherapy, psychosocial therapy, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of psoriasis vulgaris or psoriatic arthritis
* Submission of a specialist medical certificate attesting to the presence of at least one of the following ICD-10-GM diagnoses: Psoriasis vulgaris (L 40.0, L 40.7), Psoriatic arthritis (L40.5, M07.x)
* Impaired health-related quality of life (DLQI > 10)
* Consent to participate
* Sufficient understanding of the German language

Exclusion Criteria:

* Presence of another subtype of psoriasis (pustular psoriasis, guttate psoriasis, inverse psoriasis, erythrodermic psoriasis, or drug-induced psoriasis) or psoriatic arthritis without skin involvement
* Presence of malignancies
* Presence of other chronic diseases with strong negative influence on quality of life
* Currently undergoing psychiatric treatment / current presence of a severe psychiatric diagnosis
* Insufficient language and/or IT skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | 3 months
  Total score of the Dermatology Life Quality Index (DLQI). Total score ranging from 0-30; higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Psoriasis Severity | 3 months, 6 months, 12 months
  Total score of the Self-Administered Psoriasis Area Severity Index (PASI). Total score ranging from 0-72; higher scores mean a worse outcome.
Depressive Symptoms | 3 months, 6 months, 12 months
  Total score of the Patient Health Questionnaire (PHQ-9). Total score ranging from 0-27; higher scores mean a worse outcome.
Body Surface Area (BSA) | 3 months, 6 months, 12 months
  Body Surface Area (BSA) is a measure used to determine the extent of skin involvement in psoriasis. Total score ranging from 0-100; higher scores mean a worse outcome.
Health-Related Quality of Life | 6 months, 12 months
  Total score of the Dermatology Life Quality Index (DLQI). Total score ranging from 0-30; higher scores mean a worse outcome.

OTHER OUTCOMES:
Patient Activation | 3 months, 6 months, 12 months
  Total score of the Patient Activation Measure-13 (PAM-13). Total score ranging from 0-100; higher scores mean a better outcome.
Self-Esteem | 3 months, 6 months, 12 months
  Total score of the Rosenberg Self-Esteem Scale (RSE). Total score ranging from 0-30; higher scores mean a better outcome.
Body Mass Index | 3 months, 6 months, 12 months
  Body mass index (BMI) is a simple measure of body fat based on height and weight. Higher values mean a worse outcome.
Alcohol Consumption | 3 months, 6 months, 12 months
  Total score of the Alcohol use Disorders Identification Test - Consumption Items (AUDIT-C). Total score ranging from 0-12; higher scores mean a worse outcome.
Cigarette Smoking | 3 months, 6 months, 12 months
  Cigarette smoking will be assessed with a single question 'How often do you smoke cigarettes?', with response options 'Never/rarely/sometimes/often/very often', coded from 0-4. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Gieler, Prof. Dr., Principal Investigator — University of Giessen
Locations (1):
- GAIA AG, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No